CLINICAL TRIAL: NCT01528644
Title: Study to Measure the Absorption of Iron From Ferrous Gluconate Incorporated Into Alginate Beads.
Brief Title: Iron & Alginate Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BBSRC grant:BB/G0055833/1; 2011/2012-05 (Other: University of East Anglia)
Record Dates: First submitted 2012-01-17; First posted 2012-02-08 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Iron Deficiency; Anaemia
Keywords: iron; fortification; alginate; iron deficiency
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — Iron; ferrous gluconate; Capsules

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Iron in beads (Experimental): All experimental days will be exactly the same with the exception of the test meal administered to the volunteer. Volunteers will undergo a 10 hour overnight fast from 10:00pm, then they will be asked to attend the CRTU at approximately 8:00 am the following morning. A nurse will take and record the volunteer's blood pressure and if within the range an intravenous (i.v.) cannula will be inserted into a vein in one of the volunteer's arms. The cannula will remain in situ for six hours. After the first blood sample (t=0) will be taken, volunteers will consume one out of 4 test meals. After consumption further blood samples will be collected at: 20, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 min. Blood samples will subsequently be analysed for serum iron concentrations.
  Interventions: Dietary Supplement: alginate beads containing ferrous gluconate
- Iron in capsule (Experimental): All experimental days will be exactly the same with the exception of the test meal administered to the volunteer. Volunteers will undergo a 10 hour overnight fast from 10:00pm, then they will be asked to attend the CRTU at approximately 8:00 am the following morning. A nurse will take and record the volunteer's blood pressure and if within the range an intravenous (i.v.) cannula will be inserted into a vein in one of the volunteer's arms. The cannula will remain in situ for six hours. After the first blood sample (t=0) will be taken, volunteers will consume one out of 4 test meals. After consumption further blood samples will be collected at: 20, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 min. Blood samples will subsequently be analysed for serum iron concentrations.
  Interventions: Dietary Supplement: ferrous gluconate in a capsule
- Iron in beads in presence of calcium (Experimental): All experimental days will be exactly the same with the exception of the test meal administered to the volunteer. Volunteers will undergo a 10 hour overnight fast from 10:00pm, then they will be asked to attend the CRTU at approximately 8:00 am the following morning. A nurse will take and record the volunteer's blood pressure and if within the range an intravenous (i.v.) cannula will be inserted into a vein in one of the volunteer's arms. The cannula will remain in situ for six hours. After the first blood sample (t=0) will be taken, volunteers will consume one out of 4 test meals. After consumption further blood samples will be collected at: 20, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 min. Blood samples will subsequently be analysed for serum iron concentrations.
  Interventions: Dietary Supplement: alginate beads with ferrous gluconate in presence of calcium
- Iron in capsule in presence of calcium (Experimental): All experimental days will be exactly the same with the exception of the test meal administered to the volunteer. Volunteers will undergo a 10 hour overnight fast from 10:00pm, then they will be asked to attend the CRTU at approximately 8:00 am the following morning. A nurse will take and record the volunteer's blood pressure and if within the range an intravenous (i.v.) cannula will be inserted into a vein in one of the volunteer's arms. The cannula will remain in situ for six hours. After the first blood sample (t=0) will be taken, volunteers will consume one out of 4 test meals. After consumption further blood samples will be collected at: 20, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 min. Blood samples will subsequently be analysed for serum iron concentrations.
  Interventions: Dietary Supplement: ferrous gluconate in a capsule in presence of calcium

INTERVENTIONS:
Dietary Supplement: alginate beads containing ferrous gluconate — After insertion of the cannula and collection of baseline blood sample a single dose of approximately 20mg of iron as ferrous gluconate incorporated into alginate beads (approximately 22.2g)and added to cola jelly (200ml) will be given to the volunteer together with 3 placebo capsules (each containing 50mg of dextrose)and cola drink (200ml). Once consumed, further blood samples will be taken at specified time points during 6 hour cannulation time. A minimum of 7 days wash out period will take place prior next intervention.
  Other Names: iron in alginate beads
  Arms: Iron in beads
Dietary Supplement: ferrous gluconate in a capsule — After insertion of the cannula and collection of baseline blood sample a single dose of approximately 20mg of iron as ferrous gluconate in a capsule and 2 placebo capsules (each containing 50mg of dextrose) followed by a cola jelly (200ml)and cola drink (200ml) will be given to the volunteer. Once consumed, further blood samples will be taken at specified time points during 6 hour cannulation time. A minimum of 7 days wash out period will take place prior next intervention.
  Other Names: iron in capsule
  Arms: Iron in capsule
Dietary Supplement: ferrous gluconate in a capsule in presence of calcium — After insertion of the cannula and collection of baseline blood sample a single dose of approximately 20mg of iron as ferrous gluconate in a capsule together with 2 calcium capsules (each containing 300mg of calcium phosphate)followed by cola jelly (200ml) and cola drink(200ml)will be given to the volunteer . Once consumed, further blood samples will be taken at specified time points during 6 hour cannulation time. A minimum of 7 days wash out period will take place prior next intervention.
  Other Names: iron in a capsule followed by calcium phosphate
  Arms: Iron in capsule in presence of calcium
Dietary Supplement: alginate beads with ferrous gluconate in presence of calcium — After insertion of the cannula and collection of baseline blood sample a single dose of approximately 20mg of iron as ferrous gluconate incorporated into alginate beads (approximately 22.2g)and added to cola jelly (200ml) will be given to the volunteer together with 2 calcium capsules (each containing 300mg of calcium as calcium phosphate, 1 placebo capsule (containing 50mg of dextrose)and cola drink (200ml). Once consumed, further blood samples will be taken at specified time points during 6 hour cannulation time. A minimum of 7 days wash out period will take place prior next intervention.
  Other Names: iron in alginate beads in presence of calcium phosphate
  Arms: Iron in beads in presence of calcium

SUMMARY:
Iron deficiency anaemia affects around two billion people worldwide. Food fortification with iron is a realistic way to combat this problem. Water soluble forms of iron are considered to be more bioavailable than nonsoluble iron compounds. However, the former often cause sensory problems when added to foods, while the latter cause fewer problems but are not generally well absorbed and are therefore ineffective as fortificants. A potential strategy for overcoming this problem is the use of water soluble iron compounds protected by a water resistant barrier, which will prevent potential organoleptic changes within fortified foods and protect the iron (from oxidation) through the digestion process thus increasing its availability. The investigators will use alginate, in the form of alginate beads, as a protective barrier for soluble iron gluconate. It has been shown that alginates bind divalent and trivalent cations and therefore may be a useful vehicle for soluble iron compounds to fortify foods.

The aim of this project is to measure the effect of alginate on iron absorption from ferrous gluconate and assess the potential modulating effect of calcium on iron absorption in the presence and absence of alginate.

DETAILED DESCRIPTION:
This study is a randomised, single blinded, cross-over trial with participants randomly allocated into two groups: A (n= 8 volunteers) and B (n=8 volunteers). The study will include a total of four arms.

By administration of test meals #1 (iron in alginate beads) and #4 (iron in a capsule) the possible protective effect of alginate on iron absorption will be investigated. By administration of test meal #2 (iron in alginate beads + calcium capsule)and #3 (iron in a capsule + calcium in a capsule)the study will investigate whether alginates can bind calcium (a well-known iron inhibitor) in vivo, thus diminish the potential negative effect of calcium on iron absorption.

Only half (8) of the volunteers will undergo treatments including calcium. Therefore group A will undergo all 4 tests, whereas group B will undergo 2 out of 4 tests.

The four test meals will be administered a week apart following an overnight fast. On each occasion blood sampling will take place over a period of 6h with samples taken via a cannula at t=0, 20, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 min. Serum samples will be analysed for iron content allowing calculation of iron absorption.

The assumptions made for the power calculation to estimate the number of volunteers are that a difference of 2.5% in iron absorption in the presence and absence of alginate ( test meal #1 and test meal #4) will be nutritionally significant. A minimum of 12 volunteers would be required to complete the study to detect a difference of 2.5% at a significance level of 0.05 for 80% power. A minimum of 8 volunteers would be required to detect a significant difference in iron absorption of 3.3% between a test meal containing 20mg of iron as iron gluconate with calcium and a test meal containing 20mg of iron as iron gluconate with calcium and alginate beads (test meals #2 and #3). This assumes a power of 80%, a level of significance of 0.05 and standard deviation of differences (within pairs) of 2.8%

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy women (aged 18-45) or male blood donors (aged 18-65)
* Serum ferritin value of ≥15 ≤ 60µg/L
* BMI >18.5 or < 30
* Willingness to consume jelly prepared with the use of gelatine from an animal source.

Exclusion Criteria:

* Diagnosed with a long-term illness requiring active treatment, e.g. diabetes, cancer, cardiovascular disease
* Currently smoking or stopped smoking in the last 12 months
* Previous or current GI disease
* Any significant co-morbidity
* Previous GI surgery
* Blood donation within the previous 3 months assuming that volume taken is above 500ml in a 4-month period
* Blood transfusion within the last 3 months
* The results of the screening tests indicate unsuitability to take part in the study
* Related to someone in the study team i.e. spouse, partner or immediate family member
* Regular prescribed medication that may interfere with iron metabolism
* Regular use of antacids and laxatives (at least once a week)
* Women who are pregnant or less than 12 months since giving birth
* Women who are breast feeding
* Vitamin supplements with or without minerals if taken more than once a week, and unwillingness to discontinue occasional use for the duration of study
* Unwillingness to discontinue use of herbal supplements for the duration of study
* Unwillingness to consume jelly prepared with animal source gelatine
* Use of antibiotics within four weeks prior to study start Parallel participation in another study which involves dietary interventions or sampling of blood that may increase the volume taken above 500ml in a 4-month period
* Asthma requiring treatment within the last two years
* Results of clinical screening which indicate a health problem which could compromise the well-being of the volunteer if they participated or which would affect the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in iron absorption | Four weekly measurements over a period of three weeks (6h Cannulation, baseline blood sample (t=0). Test meal 1, followed by blood sample collection at 20, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 min. Removal of the cannula)
  Iron absorption (by measuring iron appearance in the serum)will be measured on four occasions with a week in between each measurement. Absorption will be assessed in response to four test meals as follows: unprotected ferrous gluconate, iron gluconate incorporated into alginate beads,ferrous gluconate incorporated into alginate beads given with calcium, and unprotected ferrous gluconate given with calcium.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Fairweather-Tait, Professor, Principal Investigator — University of East Anglia
Locations (1):
- Clinical Research and Trials Unit (CRTU)/ Norfolk and Norwich University Hospital (NNUH), Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Wawer AA, Harvey LJ, Dainty JR, Perez-Moral N, Sharp P, Fairweather-Tait SJ. Alginate inhibits iron absorption from ferrous gluconate in a randomized controlled trial and reduces iron uptake into Caco-2 cells. PLoS One. 2014 Nov 12;9(11):e112144. doi: 10.1371/journal.pone.0112144. eCollection 2014. PMID 25391138